**Document:** Informed Consent Form

**Study Title:** Angiotensin II Receptor Inhibition to Improve Microvascular Function in Women Who Have Had Preeclampsia

ро.

**NCT#** 04632589

# **Document Date(s):**

Updated and approved by IRB 7/19/2024

#### INFORMED CONSENT DOCUMENT

Project Title: Angiotensin II Receptor Inhibition to Improve Microvascular Function in Women who have had Preeclampsia

**Principal Investigator:** Anna Stanhewicz, PhD

Research Team Contact: Anna Stanhewicz, PhD

W: 319-467-1732 M: 845-551-3869 email: anna-stanhewicz@uiowa.edu

Claire Goebel (Research Associate)

W: 319-335-1914

email: claire-goebel@uiowa.edu

This consent form describes the research study to help you decide if you want to participate. This form provides important information about what you will be asked to do during the study, about the risks and benefits of the study, and about your rights as a research subject.

- If you have any questions about or do not understand something in this form, you should ask the research team for more information.
- You should discuss your participation with anyone you choose such as family or friends.
- Do not agree to participate in this study unless the research team has answered your questions and you decide that you want to be part of this study.

#### WHAT IS THE PURPOSE OF THIS STUDY?

This is a research study. We are inviting you to participate in this research study because you had a preeclamptic pregnancy in the past 5 years.

The purpose of this research study is to understand how a history of preeclampsia affects blood vessel function. Preeclampsia may cause harmful changes to blood vessels and lead to cardiovascular disease. The changes affect how the body controls blood flow. This research study looks at blood flow and how a treatment for high blood pressure, losartan, affects blood flow compared to placebo in women who had preeclampsia. We also test the stiffness of blood vessels after losartan and placebo.

This study includes the use of some research drugs in a nickel-sized area of skin on your arm (acetylcholine, L-NAME, angiotensin II, norepinephrine, and sodium nitroprusside). The drugs are not approved by the U.S. Food and Drug Administration (FDA) to treat the disease being studied in this research study. Acetylcholine, angiotensin II, norepinephrine, and sodium nitroprusside are considered investigational, which means that they have not been approved by the FDA. This study also includes the use of a study medication that is taken orally (losartan compared to placebo). Losartan is approved by the FDA to treat high blood pressure, but it is not approved by the FDA to treat blood vessels after preeclampsia. In this study losartan is compared to placebo.

# **HOW MANY PEOPLE WILL PARTICIPATE?**

Approximately 20 people will take part in this study conducted by investigators at the University of Iowa.

#### HOW LONG WILL I BE IN THIS STUDY?

If you agree to take part in this study, your involvement will last for approximately 16 weeks. During those 16 weeks you will visit the UI campus 6-7 times.

Screening visit up to 1 hour
 Pick up pretreatment 1
 Pick up 24hr BP monitor
 Study Visit 1
 up to 1 hour
 minutes
 minutes
 up to 4 hours

After study visit 1 you will have a two-week washout period where you do not take any study medications but you are still enrolled in the study.

5. Pick up pretreatment 2 15 minutes (can be completed at the end of study visit 1)

6. Pick up 24hr BP monitor7. Study Visit 215 minutesup to 4 hours

In the event of an experimental failure (e.g. equipment stops working, power outage in the building during study visit, etc) you may be asked to repeat a trial. The decision to repeat a trial is up to you. If you do repeat a trial, you will be compensated for that additional trial.

#### WHAT WILL HAPPEN DURING THIS STUDY?

Screening: The researchers and/or Clinical Research Unit (CRU) staff perform the screening. The researchers measure your height and weight, blood pressure (BP), and heart rate (HR). They measure waist circumference. You fill out a health history questionnaire. You can skip any questions that you do not want to answer. The CRU staff or approved laboratory personnel draws 50 ml (<4 Tbsp) of blood from a vein in your arm. We send some of the blood to a lab to see if the proteins, blood cells, electrolytes, kidney function, etc. are within normal levels. You submit a urine sample for a pregnancy test and provide a urine sample for the measurement of urine proteins. We will use the information collected during the screening visit to determine if you are eligible to continue in the study. After the screening visit, if you are eligible to continue in the study you begin taking the pretreatment.

<u>Pretreatments:</u> We assign one of the pretreatments (losartan or placebo) for you to take for 6 weeks. The choice of the first treatment is random. This means that whichever study treatment you receive first will be determined purely by chance, like flipping a coin. You will have a **50/50** chance of receiving any one of the study treatments first. Neither you nor the research team will know which study treatment you are receiving, but we will be able to get this information quickly if we need it to ensure your safety.

- a. The losartan dose is 50 mg/day. You take 1 pill each day for 6 weeks.
- b. You come to the lab to pick up the losartan or placebo pills. You take a urine pregnancy test. If the test is positive we do not give you the pills and you are withdrawn from the study.

- We do not want you to know the identity of the pill you are taking while you are active in the study.
   If you would like to know which treatments you received at each time, we can tell you after you complete the study.
- After 6 weeks of taking the first pretreatment, you come to the lab for the experiments described below.
- Then you take no pretreatments (washout) for at least 14 days.
- You take the second pretreatment for 6 weeks.
- After 6 weeks of taking the second pretreatment, you come to the lab to repeat the experiments described below.

**24 hour Blood Pressure Monitor:** The day before your experiment visit you wear an ambulatory blood pressure monitor on your upper arm. The monitor has a cuff that automatically inflates and contains a sensor to take a blood pressure measurement every 30 minutes during the day and once every hour overnight. You remove the monitor from your arm when the 24 hours are done. You will return the monitor to the study team when you come for your study visit.

# **Microdialysis Experiments:**

### Before you arrive:

If you have questions about the study, please contact us right away. You do not eat or drink anything containing caffeine (ex. coffee, tea, Coca Cola, chocolate) for 12 hours before the experiment and do not perform strenuous physical activity for 24 hours before the experiment.

### When you arrive:

The researchers meet you in the Clinical Research Unit of the University of Iowa Hospital or the Pharmaceutical Sciences Research Building (PSRB). We measure your blood pressure, heart rate, and oral temperature. You provide a urine sample for the measurement of urine proteins. A CRU nurse or approved laboratory personnel draws your blood. Then, the rest of the study visit occurs in 118 PSRB for the intradermal microdialysis experiment.

#### **Measurements:**

Blood Pressure, Heart Rate: We measure blood pressure and heart rate throughout the experiment. We apply three sticky tabs to the skin of your chest. The tabs connect to an ECG machine that records heart rate. During the experiment, we can measure blood pressure in any of two ways. a) We inflate a cuff on your upper arm while we listen at the inside of your elbow with a stethoscope. b) Likewise, an automated machine inflates a cuff on the upper arm and uses a sensor in the cuff to measure blood pressure.

Skin Blood Flow, Skin Temperature: We measure skin blood flow and skin temperature throughout the experiment. We tape a thin probe and its holder over five sites on your forearm. The thin probe measures skin blood flow with a weak laser light. The holders measure skin temperature. We control the temperature of the holders. The holders start at 34°C (93°F). At the end of the study, we increase the temperature of the holders from 34°C to 43°C (108°F).

<u>Pulse Wave Velocity</u>: We measure the stiffness of your blood vessels by measuring how fast the pulse of blood from each heartbeat travels through your vessels. The researcher uses a small

handheld probe placed on the surface of the skin to measure your pulse at your carotid artery (on your neck), your brachial artery (near your elbow), and your femoral artery (near your thigh). We record these pulses for 20 seconds.

#### **Microdialysis (MD):**

Overview: MD involves placing very thin plastic tubing between the layers of your skin. The largest part of the tubing is about 6 times the diameter of a human hair. We pump fluid like that found in your body's tissues (lactated Ringer's solution) through the thin tubing. Lactated Ringer's solution is a fluid commonly used in hospital and healthcare settings in IVs. It is used to treat dehydration and restore fluid balance in the body.

The thin tubing acts like the very small blood vessels in your skin. There is an exchange of substances between the fluid in the tubing and the fluid in the surrounding tissue. During the experiment, we add substances to the fluid in the tubing. The substances can only reach a 2.5 cm<sup>2</sup> (0.4 inch<sup>2</sup>), nickel-sized area of skin.

MD Probe Insertion: We place a tight band around your arm so we can easily see your veins. For each MD site, we make pairs of pen-marks 2.5 cm (1 inch) apart and away from veins. The MD tubing enters and exits your skin at the marks. We remove the tight band. We clean your arm with an orange-colored fluid and alcohol. We place an ice bag on your arm for 5 minutes to numb your skin. Then we insert a thin needle into your skin at each entry mark. The needle's tip travels between the layers of skin for 2.5 cm (1 inch). It leaves your skin at the matching exit mark. We thread the MD tubing through the needle. Next, we withdraw the needle, leaving the tubing in your skin. We prepare all MD sites in this manner. Any redness of your skin subsides in about 60 - 120 minutes.

# Microdialysis Experiment Protocol (described below):

Summary: We prepare 4 MD sites as described above. At first, we record baseline measurements for all 4 sites (20 minutes). After we have collected baseline data, we change the fluid flowing through each microdialysis fiber at 5-minute intervals. We do not collect any samples from the probes. After the last amounts of acetylcholine, angiotensin II, and norepinephrine have been added, we change the fluid flowing through the tubing to lactated Ringers and warm the temperature controllers to 43°C (108°F). After 40 minutes of heating, we add SNP to the fluid in sites 1 and 2 for 5 minutes. At the end of the protocol, we remove the probes and apply a sterile dressing. If you want, we can place a bag of ice on your arm for 10 minutes to reduce any bruising that may occur. We remove all instrumentation and measure your heart rate and blood pressure before you leave.

The 4 MD sites are:

Acetylcholine Dose Response: Probe 1. Lactated Ringer's only

Probe 2. Lactated Ringer's + L-NAME

Angiotensin II Dose Response: Probe 3. Lactated Ringer's only Norepinephrine Dose Response: Probe 4. Lactated Ringer's only

## Tissue/Blood/Data Storage for Future Use

As part of this study, we are obtaining blood samples and peripheral blood mononuclear cells (white blood cells circulating in your blood) from you. We would like to study your blood samples and

mononuclear cells in the future, after this study is over. Your sample, information, and/or data may be placed in a central repository or other national repositories sponsored by the National Institutes of Health or other Federal agencies. If this happens, it will be stripped of identifiers (such as name, date of birth, address, etc). Other qualified researchers who obtain proper permission may gain access to your sample and/or data for use in approved research studies that may or may not be related to the purpose of this study. The use of the blood and mononuclear cells *will not* include whole genome sequencing as part of future use.

The tests we might want to use to study your blood and mononuclear cells may not even exist at this time. Therefore, we are asking for your permission to store your blood and mononuclear cells so that we can study them in the future. These future studies may provide additional information that will be helpful in understanding preeclampsia and cardiovascular disease, but it is unlikely that what we learn from these studies will have a direct benefit to you. It is possible that your blood and mononuclear cells might be used to develop products, tests, or discoveries that could be patented and licensed. In some instances, these may have potential commercial value and may be developed by the Investigators, University of Iowa, commercial companies, organizations funding this research, or others that may not be working directly with this research team. However, donors of blood and mononuclear cells do not retain any property rights to the materials. Therefore, there are no plans to provide financial compensation to you should this occur.

Your blood and mononuclear cells will be stored with a code which may be linked to your name and date of birth. If you agree now to future use of your blood and mononuclear cells but decide in the future that you would like to have it removed from future research, you should contact Anna Stanhewicz (319-467-1732, anna-stanhewicz@uiowa.edu). However, if some research with your blood and mononuclear cells has already been completed, the information from that research may still be used.

Please place your initials in the blank next to Yes or No for each of the questions below:

| My blood and mononuclear cells may be stored/shared for future research in cardiovascular disease and preeclampsia | | | | |
|---|---|---|---|---|
| Yes | No | | | |
| My blood an | d mononuclear cells | s may be stored/share | d for future research | h for any other purpose. |
| Yes | No | | | |

### WILL I BE NOTIFIED IF MY STUDY VISIT RESULT(S) IN AN UNEXPECTED FINDING?

The results from the skin blood flow data we collect in this research study are not the same quality as what you would receive as part of your routine health care. The results will not be reviewed by a physician. Due to this, you will not be informed of any unexpected findings. The results of your study visit will not be placed in your medical record with your primary care physician or otherwise. If you believe you are having symptoms that may require care, you should contact your primary care physician.

If you consent, we may contact you to participate in future studies with our laboratory group. We will

keep your name, race/ethnicity, age, pregnancy history, and contact information for this purpose. Participating in this study does not mean that you are obligated to participate in any future studies. A separate consent document would be signed for future studies.

May we keep your name, race/ethnicity, age, pregnancy history, and contact info to contact you for future studies? Please place your initials in the blank next to Yes or No for each of the questions below:

| Yes |
|--------|
| <br>No |

#### WHAT ARE THE RISKS OF THIS STUDY?

You may experience one or more of the risks indicated below from being in this study. In addition to these, there may be other unknown risks, or risks that we did not anticipate, associated with being in this study.

**Losartan:** Losartan is a blood pressure lowering medication, that is commonly prescribed to lower blood pressure in people who have high blood pressure. It is also used to treat diabetic kidney disease. Losartan is part of a group of drugs called "angiotensin receptor blockers (ARBs)". You will not be included in this study if you have an allergy to losartan. You could have an allergy that is unknown to you. An allergic reaction could include hives, difficult breathing, and swelling of your face, lips, tongue, or throat. Losartan can cause harm or death to an unborn baby. Because of this, women enrolled in this study will be required to use an effective form of birth control. Effective forms of birth control are:

- hormonal patch, implant or pill;
- intrauterine device;
- consistent use of barrier contraceptive;
- prior medical procedure to prevent pregnancy (e.g. tubal ligation, or vasectomy in current partner)

You will be excluded from this study if you are pregnant or planning to become pregnant within the next 6 months. We will perform a urine pregnancy test when we give you the medication to check that you are not pregnant. If you suspect that you have become pregnant while you are in this study, stop taking the medication immediately and notify the researchers.

Please tell us if you have any side effects of the medication including the following side effects.

#### Less serious side effects:

- "colds" (upper respiratory infection)
- · mild dizziness
- stuffy nose
- back pain
- diarrhea

#### Serious side effects:

- Allergic reaction. Symptoms of an allergic reaction are swelling of the face, lips, throat or tongue.
- Low blood pressure (hypotension)
- Swelling in feet, ankles, or hands, or unexplained weight gain.

Microdialysis: The risks are less than that for a blood draw because microdialysis uses only a small, local area of skin. In contrast, a blood draw involves not only skin, but also large blood vessels and blood. You are likely to have some pain and bruising like that from a blood draw. However, we use ice to numb your arm when we insert the tubing. Also, we use a small needle, which is less painful than a typical needle for drawing blood, when we insert the tubing. You are not likely to have pain after the tubing is in place. You may feel a little pain when we remove the tubing from your skin. Needles make some people feel lightheaded or cause them to faint. Although rare, the tubing could break as we remove it from the skin. Then we remove the tubing still in your skin by pulling on the other end of it. This presents no added risk for you. Even more rare, the tubing could break so that a piece of the tubing is left under your skin. In this case, we treat any tubing still in your skin like a splinter. We stop any mild bleeding with mild pressure and sterile gauze. Infection is possible. We keep the risk of infection very small by using sterile techniques and supplies like those used with blood draws. We apply a sterile bandage to the site after the experiment. We tell you how to take care of the site.

Fluid flowing through the tubing: The substances flowing through the tubing only go to a 2.5 cm<sup>2</sup> (0.4 inch<sup>2</sup>) area of skin at each tubing site. The amount that enters the skin is very small. However, there is a chance of having a bad reaction to the substances. This reaction could produce redness, itching, rash, and/or swelling. A worse reaction could also cause fever, breathing problems, changes in pulse, convulsions, and/or fainting. We and other researchers have used these substances with microdialysis in skin. There have been no reports that these substances caused bad reactions. If a bad reaction should occur, we summon medical help.

Lactated Ringer's Solution: This fluid is similar to the natural fluids in your skin. This fluid contains salt, potassium, lactate, and chloride. The acid content is like that in your body's natural fluids. A bad reaction to this fluid is highly unlikely.

Acetylcholine, Angiotensin II, Norepinephrine, L-NAME, SNP: These substances stop or mimic the action of your body's natural chemicals upon the blood vessels in the skin. A small amount of these substances enter the skin around the tubing. This only affects the blood flow in the vessels in that nickel-sized area of skin. The effect of these substances in your skin is gone within an hour after the experiment.

Acetylcholine (ACh) - causes blood vessels to dilate (get wider).

Angiotensin II (Ang II) - causes blood vessels to constrict (get smaller).

L-NAME – like a substance made by your body; prevents some blood vessel dilation.

Norepinephrine – causes blood vessels to constrict (get smaller)

Sodium Nitroprusside (SNP) - causes blood vessels to dilate as much as they can.

**Laser Doppler Flowmetry:** We use a weak laser light at each microdialysis site to measure your skin's blood flow. The weak lasers can hurt your eye if you stare into the light for a long time. We do not turn on the laser until the probes are taped to a surface. The tape may irritate your skin.

**Blood Pressure:** The researchers measure blood pressure with the method used in a doctor's office and they can use a machine. A cuff inflates on the upper arm. As the cuff slowly deflates, the researchers listen with a stethoscope at the bend in the elbow or the machine takes a reading. During the short time the researchers inflate the cuff, your arm may feel numb or tingly. The cuff could cause mild bruising.

**Povidone Iodine:** Researchers and hospitals use this orange-colored fluid to clean the skin. You could have a bad reaction if you are allergic to iodine. You need to inform us if you have this allergy. In this case, we use only alcohol instead. A bad reaction could cause redness, itching, rash, and/or swelling. A worse reaction could also cause fever, breathing problems, changes in pulse, convulsions, and/or fainting.

**Blood Draw**: Blood draws often cause mild pain, bruising, swelling, or bleeding. There is also a slight chance of infection or a small clot. If you are nervous about needles, blood pressure and heart rate may increase for a little while. You may also feel lightheaded, sick to your stomach, or may faint. Using the same techniques used in hospitals keeps the chance of infection minimal.

**Tape and sticky disks:** The tape or sticky disks could cause a rash. During screening, you tell us if you are sensitive to tape. If a disk sticks very strongly, removing the disk could cause an abrasion like a rug-burn on your skin. An abrasion can feel tender or slightly painful, and can increase risk of infection. If you are sensitive to tape, you may have an increased chance for abrasion. If you get an abrasion, antibiotic ointment and a sterile bandage are applied. We tell you how to take care of the site.

**Medical Screening:** You may feel shy about giving health information. The staff collects the information in a private and professional manner. You may feel shy about being measured. You may request someone of the same sex to conduct the screening.

**Initial screening form:** Only members of our lab group use this form. We use the form to help decide whether you are a good candidate for the study. You may feel shy about answering questions. You may request someone of the same sex to ask you the questions. We collect the information in a private and professional manner. We keep the completed form confidential and secure.

**ECG Heart Rate:** This machine measures the electrical activity of your heart. You have 3 wires from the machine taped to spots on your chest. There have been no adverse effects. The tape may irritate.

**Local heating:** We measure the temperature of your skin under the holders. During heating, the skin feels very warm but will not hurt. The heating makes the skin under the holder red like when you take a hot bath. The redness goes away within several hours. Some people may be more sensitive to heating. If your arm feels too hot, tell us, and we will reduce or stop the heating.

**Latex:** Some gloves and medical materials are made of latex rubber. You will inform us if you are allergic to latex and decline to participate in the study.

There is a risk of loss of confidentiality if your information or your identity is obtained by someone other than the investigators, but precautions will be taken to prevent this from happening. The confidentiality of your electronic data created by you or by the researchers will be maintained to the degree permitted by the technology used. Absolute confidentiality cannot be guaranteed.

#### WHAT ARE THE BENEFITS OF THIS STUDY?

We don't know if you will benefit from being in this study.

However, we hope that, in the future, other people might benefit from this study because an understanding of blood flow in women who have had preeclampsia may help us to better understand the connection between preeclampsia and cardiovascular disease. This knowledge could aid the development of new methods for managing the risks in these women.

### WILL IT COST ME ANYTHING TO BE IN THIS STUDY?

You will not have any costs for being in this research study. You/your insurance company will remain responsible for your regular clinical care.

### WILL I BE PAID FOR PARTICIPATING?

You will be paid for being in this research study. You may need to provide your address if a check will be mailed to you.

**Pre-treatment**: \$30 per treatment (\$5/week for 6 weeks)

**24-hour blood pressure monitor**: \$10

Experimental visits: \$100 per visit (\$15/microdialysis probe + \$10 for pulse wave velocity

measurements + \$7.50/hour for completing the experiment)

Total for completing the study: \$280 (two pre-treatment periods, two 24 hour blood pressure monitors,

two completed study visits)

You will be given a parking pass for time involved at study and screening visits.

Pro-rating: Subjects can receive payment for pre-treatment and experiments that are partially completed. The researchers pay an amount of money equal to the part completed. For instance, if a subject completes half of Experiment 1, the subject receives \$15.00 for each probe inserted plus \$7.50 for each hour they completed. The researchers may ask subjects to repeat a trial. If subjects agree to repeat a trial, they receive payment for the repeated trial as stated above.

#### WHO IS FUNDING THIS STUDY?

The University and the research team are receiving no payments from other agencies, organizations, or companies to conduct this research study.

# WHAT IF I AM INJURED AS A RESULT OF THIS STUDY?

- If you are injured or become ill from taking part in this study, medical treatment is available at the University of Iowa Hospitals and Clinics.
- The University of Iowa does not plan to provide free medical care or payment for treatment of any illness or injury resulting from this study unless it is the direct result of proven negligence by a University employee.
- If you experience a research-related illness or injury, you and/or your medical or hospital insurance carrier will be responsible for the cost of treatment.

#### WHAT ABOUT CONFIDENTIALITY?

It is possible that other people such as those indicated below may become aware of your participation in this study and may inspect and copy records pertaining to this research. Some of these records could contain information that personally identifies you.

- federal government regulatory agencies,
- U.S. Food and Drug Administration
- National Institutes of Health
- auditing departments of the University of Iowa, and
- the University of Iowa Institutional Review Board (a committee that reviews and approves research studies)

To help protect your confidentiality, we will limit the use and sharing of your personal research information to people who have a need to review this information. We keep the list that matches your name with your code number in a locked file or password protected file on a computer in a room that is locked when unoccupied. Only authorized members of the lab have access to the list. We label your research records with your code number and keep them in a locked file or password protected computer in a room that is locked when unoccupied. We label your research samples with your code number only. If we write a report or article about this study or share the study data set with others, we will do so in such a way that you cannot be directly identified.

The University of Iowa Hospitals and Clinics generally requires that we document your participation in research occurring in a University of Iowa Health Care facility. This documentation will be in either your medical record or a database maintained on behalf of the institution reflecting that you are participating in this study. The information included will provide contact information for the research team as well as information about the risks associated with this study. We will keep this Informed Consent Document in our research files; it will not be placed in your medical record chart.

If we write a report or article about this study or share the study data set with others, we will do so in such a way that you cannot be directly identified.

To further protect your privacy, the researchers have obtained a Certificate of Confidentiality from the Department of Health and Human Services (DHHS). This Certificate means that the researchers cannot be forced (for example by court subpoena) to disclose information that may identify you in any federal, state, or local civil, criminal, administrative, legislative, or other proceeding. However, a Certificate of Confidentiality does not prohibit the researcher from disclosing information about you or your involvement in this research that you have agreed to disclose or make available. For example, if you request in writing that information about you or your participation in the research be released to an insurance company, the researcher may not use the Certificate of Confidentiality to withhold this information. This means that you and your family should actively protect your own privacy. Finally, the researcher is not prevented from taking steps, including reporting to appropriate authorities, to prevent serious harm to yourself or others. You may receive a copy of the Certificate of Confidentiality upon request.

### WILL MY HEALTH INFORMATION BE USED DURING THIS STUDY?

The Federal Health Insurance Portability and Accountability Act (HIPAA) requires University of Iowa Health Care to obtain your permission for the research team to access or create "protected health information" about you for purposes of this research study. Protected health information is information that personally identifies you and relates to your past, present, or future physical or mental health condition or care. We will access or create health information about you, as described in this document, for purposes of this research study. Once University of Iowa Health Care has disclosed your protected health information to us, it may no longer be protected by the Federal HIPAA privacy regulations, but we will continue to protect your confidentiality as described under "Confidentiality."

We may share your health information related to this study with other parties including federal government regulatory agencies, the University of Iowa Institutional Review Boards and support staff, the National Institutes of Health, and the U.S. Food and Drug Administration.

You cannot participate in this study unless you permit us to use your protected health information. If you choose *not* to allow us to use your protected health information, we will discuss any non-research alternatives available to you. Your decision will not affect your right to medical care that is not research-related. Your signature on this Consent Document authorizes University of Iowa Health Care to give us permission to use or create health information about you.

Although you may not be allowed to see study information until after this study is over, you may be given access to your health care records by contacting your health care provider. Your permission for us to access or create protected health information about you for purposes of this study has no expiration date. You may withdraw your permission for us to use your health information for this research study by sending a written notice to: Anna Stanhewicz, 410 Field House, 225 South Grand Avenue, Iowa City, IA 52242. However, we may still use your health information that was collected before withdrawing your permission. Also, if we have sent your health information to a third party, such as the study sponsor, or we have removed your identifying information, it may not be possible to prevent its future use. You will receive a copy of this signed document.

# **IS BEING IN THIS STUDY VOLUNTARY?**

Taking part in this research study is completely voluntary. You may choose not to take part at all. If you decide to be in this study, you may stop participating at any time. If you decide not to be in this study, or if you stop participating at any time, you won't be penalized or lose any benefits for which you otherwise qualify.

### Will I Receive New Information About the Study while Participating?

If we obtain any new information during this study that might affect your willingness to continue participating in the study, we'll promptly provide you with that information.

# Can Someone Else End my Participation in this Study?

Under certain circumstances, the researchers might decide to end your participation in this research study earlier than planned. This might happen if you become pregnant, if the researcher decides to end the study early, or if for any reason the researcher decides that it is no longer safe for you to continue.

#### WHAT IF I HAVE QUESTIONS?

We encourage you to ask questions. If you have any questions about the research study itself, please contact: Anna Stanhewicz (319)467-1732 or Claire Goebel (319)335-1914. If you experience a research-related injury, please contact: Anna Stanhewicz (319)467-1739.

If you have questions, concerns, or complaints about your rights as a research subject or about research related injury, please contact the Human Subjects Office, 105 Hardin Library for the Health Sciences, 600 Newton Rd, The University of Iowa, Iowa City, IA 52242-1098, (319) 335-6564, or e-mail <a href="mailto:irb@uiowa.edu">irb@uiowa.edu</a>. General information about being a research subject can be found by clicking "Info for Public" on the Human Subjects Office web site, <a href="http://hso.research.uiowa.edu/">http://hso.research.uiowa.edu/</a>. To offer input about your experiences as a research subject or to speak to someone other than the research staff, call the Human Subjects Office at the number above.

| This Informed Consent Document is not a contract. It is a valuring the study if you decide to participate. You are not was Informed Consent Document. Your signature indicates that you, that your questions have been answered, and that you receive a copy of this form. | raiving any legal rights by signing this this research study has been explained to |
|---|---|
| Subject's Name (printed): | |
| (Signature of Subject) | (Date) |
| Statement of Person Who Obtained Consent | |
| I have discussed the above points with the subject or, where appropriate, with the subject's legally authorized representative. It is my opinion that the subject understands the risks, benefits, and procedures involved with participation in this research study. | |
| (Signature of Person who Obtained Consent) | (Date) |